CLINICAL TRIAL: NCT04205682
Title: A Randomised Controlled Trial of Cannabidiol (CBD) for the Treatment of Alcohol Withdrawal
Brief Title: Cannabidiol (CBD) for the Treatment of Alcohol Withdrawal
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: South West Sydney Local Health District (Other)
Collaborators: University of Sydney (Other); South Eastern Sydney Local Health District (Other Government)
Responsible Party: Principal Investigator, Professor Paul Haber, Director, South West Sydney Local Health District
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: X18-0163
Record Dates: First submitted 2019-11-05; First posted 2019-12-19 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Alcohol Withdrawal; Alcohol Dependence
MeSH Terms: conditions — Alcoholism | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cannabidiol (CBD) (Experimental): Drug: Cannabidiol (day 1: 1200 mg (800 mg BD); day 2-4: 800 mg (400 mg BD); day 5: placebo BD).
  Interventions: Drug: Cannabidiol
- Placebo (Placebo Comparator): Drug: Placebo (days 1-5: placebo matched BD)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cannabidiol — CBD capsules administered BD for 4-days (800-1200 mg/day), placebo day 5
  Arms: Cannabidiol (CBD)
Drug: Placebo — Placebo capsules administered BD for 5 days
  Arms: Placebo

SUMMARY:
This study will explore the effectiveness and tolerability of Cannabidiol (CBD) in the treatment of alcohol withdrawal symptoms in an inpatient setting, in a double-blind randomised placebo-controlled trial.

DETAILED DESCRIPTION:
New treatment strategies for treating symptoms of alcohol dependence are urgently needed. Although alcohol related disorders are a leading cause of preventable death in Australia, their treatment is generally not evidence-based. Contemporary treatment for managing alcohol withdrawal in Australia involves administration of benzodiazepines that, while often effective for managing withdrawal symptoms, have concerns regarding their use including: a major abuse liability potential in this population; their sedating effects and potential for adverse events (e.g. falls, overdose, cognitive impairment) if used in combination with other sedatives; and an increased risk of relapse due to symptoms of alcohol dependence that return after cessation of treatment (e.g. increased sleep problems and anxiety). However, no other safe and effective alternatives to benzodiazepines in treating alcohol withdrawal have yet been demonstrated.

This project will pilot the clinical efficacy and tolerability of Cannabidiol (CBD) relative to placebo in the treatment of alcohol withdrawal in an inpatient setting across two study sites.

This is a double-blind, randomised controlled design. The trial will recruit 52 participants undergoing alcohol withdrawal, using a 1:1 random allocation into one of two treatment groups as follows: (1) CBD (Day 1: 1200 mg/day; Day 2-4: 800 mg/day; Day 5: placebo washout; n = 26), or (2) matched placebo (n = 26). All participants will be administered a symptom triggered diazepam medication regimen, as per conventional best-practice management of alcohol withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years;
* At least one prior episode 2 days or longer in duration during which the participant experienced withdrawal symptoms that caused significant incapacitation (e.g. inability to work or do normal activities) OR at least one prior inpatient or outpatient medical detoxification during which the participant exhibited withdrawal symptoms of significant magnitude that sedative-hypnotic or anticonvulsant medication was required at least once on 2 consecutive days after cessation of or reduction in the use of alcohol following 2 weeks or more of heavy daily consumption;
* Average consumption of at least 8 standard drinks per day for at least 2 weeks prior to enrolment in the study;
* Adequate cognition and English language skills to give valid consent and complete research interviews;
* Willingness to give written informed consent

Exclusion Criteria:

* Treatment/ingestion during the previous week of benzodiazepines or other sedative-hypnotic medications or history of recent chronic treatment with sedative-hypnotic medication as evidenced by a negative urine drug screen at baseline
* History of alcohol withdrawal related seizures
* Substance use in the previous week, defined as > 3 times per week (not including nicotine or caffeine), inclusive of non-prescribed pharmaceuticals (ATOP to be collected at screening)
* Active major psychiatric disorder associated with psychosis, or significant suicide risk (e.g. Bipolar, Schizophrenia)
* Pregnancy or lactation - Women shall be advised to use reliable contraception for the duration of drug therapy and a urine pregnancy test will be performed where necessary
* History of confirmed seizures during adulthood, and/or current use of anti-epileptic drugs (AED)
* Diagnosis of epilepsy, and/or current use of anti-epileptic drugs (AED)
* Serious medical illness impacting on safety/participation, defined as an unstable medical state in the opinion of the trial medical officer
* Low body weight (body mass index < 17)
* Severe cognitive impairment or insufficient English or literacy to complete study processes
* Concurrent use of drugs potentially exacerbated by CBD via CYP3A5

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Diazepam | 5 day admission period
  Diazepam use over the 5-day withdrawal period (which due to symptom triggered regimen is a proxy measure for withdrawal severity). Measured by total diazepam use over 5 day period.

SECONDARY OUTCOMES:
Alcohol Withdrawal Severity | 5 day admission period
  Measured by Alcohol Withdrawal Scale (AWS), minimum score is 0, maximum score is 27 where higher scores indicate greater withdrawal severity.
Self-reported Alcohol Withdrawal Severity | 5 day admission period (twice daily)
  As measured by the Alcohol Withdrawal Severity Checklist (AWSC), a self-report measure of withdrawal severity, minimum score is 0, maximum score is 64 where higher scores indicate greater self-reported withdrawal severity.
Self-reported alcohol craving | Baseline, Day 5, and Day 12 and 33 Follow Up
  As measured by the Penn Alcohol Craving Scale (PACS), minimum score is 0, maximum score is 30 where higher scores indicate greater alcohol craving
Self-reported urges to drink | Twice Daily, days 1-5
  As measured by the Alcohol Urge Questionnaire (AUQ), minimum score is 8, maximum score is 56, where higher scores indicate greater urges to drink
Actiwatch for sleep quality | 5 day admission period
  as measured using data obtained from the actiwatch worn by participants for duration of inpatient stay
Self-reported sleep quality | Baseline, Day 5, and Follow Up (Day 12, Day 33)
  as measured using the Insomnia Severity Index (ISI), minimum score is 0, maximum score is 28, where higher scores indicate greater insomnia severity.
Subjective measure of patient satisfaction | Day 5 and follow up (day 12 and 33)
  Measured using the Treatment Satisfaction Questionnaire for Medication (TSQM), minimum score is 13, maximum score is 80, where higher scores indicate greater treatment satisfaction.
Liver function tests for clinical markers of liver injury | Baseline and follow up (day 12 and 33).
  as measured by levels of liver enzymes, Alanine Transaminase (ALT), Alkaline Phosphatase (ALP) and Aspartate Transaminase (AST) in blood
Plasma levels of benzodiazepines | Daily (days 1-5)
  As measured by concentration of benzodiazepines in blood plasma
Plasma levels of cannabidiol | Daily (days 1-5)
  As measured by concentration of cannabidiol in blood plasma
Mood | Baseline, day 5 and follow up day 12 and 33.
  Depression, Anxiety and Stress Symptoms measured by the Depression, Anxiety and Stress Scale (DASS-21), minimum score is 0, maximum score is 63, where higher scores indicate greater levels of depression, anxiety and stress.
Cognitive Functioning | Baseline, day 5 and follow up day 12 and 33.
  As measured by the Montreal Cognitive Assessment (MoCA), maximum score is 30 and where higher scores indicate greater cognitive functioning.
Cognitive Functioning | Baseline, day 5 and follow up day 12 and 33.
  Executive functioning measured by time taken to complete the Trail Making Test A and B (in seconds), where lower scores indicate greater functioning.
Comorbid Anxiety Disorders | 4 week follow up (day 33)
  Assessed using the MINI Neuropsychiatric Interview indicating the presence or absence of anxiety disorders

CONTACTS AND LOCATIONS:
Overall Officials: Paul Haber, MBBS, Principal Investigator — Sydney Local Health District; Nicholas Lintzeris, MBBS, Principal Investigator — South Eastern Sydney Local Health District; Iain McGregor, PhD, Principal Investigator — University of Sydney; Kirsten Morley, PhD, Principal Investigator — University of Sydney
Locations (2):
- Australia (2):
  - Sydney and Sydney Eye Hospital, Sydney, New South Wales
  - Royal Prince Alfred Hospital, Sydney, New South Wales